CLINICAL TRIAL: NCT00359047
Title: Recognizing Osteoporosis and Its Consequences in Quebec (ROCQ) Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry); Sanofi (Industry); Procter and Gamble (Industry); Amgen (Industry); Eli Lilly and Company (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Jacques Brown, Clinical researcher, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUL 61.05.05
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Fragility fracture; Women; Randomised control trial; Patient education; Diagnosis; Treatment
MeSH Terms: conditions — Osteoporosis; Disease | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Documentation (Experimental): Written educational material on osteoporosis for the participant and the physician.
  Interventions: Behavioral: Documentation
- Video (Experimental): A 15-minute educational video on osteoporosis as well as written documentation on osteoporosis for the participant and the physician.
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Documentation — Participants will receive written educational material for themselves as well as the Guidelines document for their physician (same written material as in the Educational Video Group). They will be asked to revisit their physician and provide written documentation inviting him/her to consider a complementary investigation and an adequate treatment according to the 2002 Clinical Practice Guidelines for the Diagnosis and Management of Osteoporosis in Canada
  Arms: Documentation
Behavioral: Video — Participants will receive a 15-minute educational video on osteoporosis. They will also receive written educational material for themselves and a Guidelines document for their physician. They will be asked to revisit their physician and provide the written documentation inviting her/him to consider a complementary investigation and an adequate treatment according to the 2002 Clinical Practice Guidelines for the Diagnosis and Management of Osteoporosis in Canada. Should participants wish to obtain additional information on osteoporosis, they will be provided with a toll-free number (1-866-571-ROCQ) to contact
  Arms: Video

SUMMARY:
The aim of the ROCQ programme is to improve the use of evidence based osteoporosis diagnostic and treatment strategies for women 50 years and over who have suffered a fragility fracture. This objective will be achieved by concentrating on a realistic evaluation of the present diagnosis and treatment rate of osteoporosis following a fragility fracture and comparing it to an optimal situation (care gap) and proposing interventions that promote new approaches to treating osteoporosis by health professionals as well as providing targeted interventions for the patient. The efficacy of these interventions will be evaluated using a randomized control design.

DETAILED DESCRIPTION:
ROCQ is a patient health-management programme and prospective cohort study. Within the ROCQ programme, educational interventions to improve osteoporosis management will be evaluated using a randomized-control design. The programme is composed of a promotional campaign, three main phases and a 20-year follow-up.

At phase 1, 0 to 16 weeks after the fracture, participants with fragility and traumatic fractures will be recruited and will be asked information regarding their fracture.

At phase 2, 6 to 8 months after the fracture, all participants will complete questionnaires to evaluate demographic and clinical features, risk factors for osteoporosis, co-morbidities, status of diagnosis and treatment, and the EQ-5D. The current medical management of osteoporosis (or the care gap in diagnosis and treatment) will be measured using this questionnaire at phase 2. Once the phase 2 questionnaire has been completed, Only participants with fragility fractures will be randomized to one of the three following educational intervention groups: 1) the Educational Video Group, 2) the Documentation Group, or 3) the Control Group.

At phase 3, 12 to 14 months after randomization, the effectiveness of the interventions will be assessed by re-administering the questionnaires to participants who experienced a fragility fracture at baseline. The questionnaires evaluate the status of diagnosis and treatment of osteoporosis, modifiable risk factors and the health-related quality of life (EQ-5D). The impact of the interventions on the participants will be assessed by comparing diagnosis and treatments rates in each intervention arm.

If the long-term viability of the programme is secured, participants with fragility and traumatic fractures will be followed for a maximum period of 20 years using specific encoded personal data contained in the RAMQ and Quebec's drug plan databases.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 50 years and over.
* Not residing in a long-term care hospital before the fracture.
* Able to understand the programme information and consent form.
* Must voluntarily accept to participate in this programme and sign the consent form.
* Participants must have a fragility or traumatic fracture of one of the following sites: wrist, forearm, humerus, scapula, clavicle, sternum, thoracic or lumbar vertebrae, pelvis, sacrum, hip, femur, proximal and distal tibia, fibula (including ankle), and foot.
* Participants must be able to answer the questionnaires via phone interviews

Exclusion Criteria:

* Unable to understand the purpose of the programme.
* Participants with a traumatic fracture of one of the following sites: cervical, skull and face, hand and finger, toe, metatarsus, and patella.
* Pathological fracture.
* Women currently participating in a clinical trial requiring them to take a medication for osteoporosis.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2830 (Actual)
Dates: Start 2003-06; Primary Completion 2007-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The present diagnostic and treatment rates of osteoporosis 6 months after a fragility fracture | June 2007
The osteoporosis diagnostic rate and on the osteoporosis pharmacological treatment rate 12 months after the educational interventions | June 2007
The average 5-year, 10-year, 15-year, and 20-year probabilities of a fragility fracture by age, site of previous fragility fracture, and type of ROCQ intervention. | July 2009

SECONDARY OUTCOMES:
Changes of modifiable risk factors for osteoporosis 12 months after the intervention | September 2009
Proportion of fragility versus traumatic fractures. | June 2007
Health care resource utilization associated with specific types of fragility fracture and recurrent fractures. | September 2010
Assess health utility index (EQ-5D) after a fragility fracture. | September 2010
Satisfaction with the process of care before and after implementing ROCQ's interventions. | June 2010
One-year mortality rate following a fragility fracture. | May 2009
Persistence to pharmacological treatment 12 months after the intervention | October 2009
Incidence of recurrent fracture and health care resources utilization between women who previously had a fragility fracture and those who had a traumatic fracture. | November 2010

CONTACTS AND LOCATIONS:
Overall Officials: Jacques P Brown, MD, Principal Investigator — CHU de Quebec
Locations (1):
- CHUdeQuebec, CHUL, Québec, Quebec, Canada

REFERENCES:
- [Background] Bessette L, Ste-Marie LG, Jean S, Davison KS, Beaulieu M, Baranci M, Bessant J, Brown JP. Recognizing osteoporosis and its consequences in Quebec (ROCQ): background, rationale, and methods of an anti-fracture patient health-management programme. Contemp Clin Trials. 2008 Mar;29(2):194-210. doi: 10.1016/j.cct.2007.07.007. Epub 2007 Jul 24. PMID 17766187
- [Result] Bessette L, Jean S, Davison KS, Roy S, Ste-Marie LG, Brown JP. Factors influencing the treatment of osteoporosis following fragility fracture. Osteoporos Int. 2009 Nov;20(11):1911-9. doi: 10.1007/s00198-009-0898-x. Epub 2009 Mar 31. PMID 19333675
- [Result] Beaudoin C, Bessette L, Jean S, Ste-Marie LG, Brown JP. The impact of educational interventions on modifiable risk factors for osteoporosis after a fragility fracture. Osteoporos Int. 2014 Jul;25(7):1821-30. doi: 10.1007/s00198-014-2618-4. Epub 2014 Feb 12. PMID 24519745
- [Result] Bessette L, Jean S, Lapointe-Garant MP, Belzile EL, Davison KS, Ste-Marie LG, Brown JP. Direct medical costs attributable to peripheral fractures in Canadian post-menopausal women. Osteoporos Int. 2012 Jun;23(6):1757-68. doi: 10.1007/s00198-011-1785-9. Epub 2011 Sep 17. PMID 21927921
- [Result] Bessette L, Davison KS, Jean S, Roy S, Ste-Marie LG, Brown JP. The impact of two educational interventions on osteoporosis diagnosis and treatment after fragility fracture: a population-based randomized controlled trial. Osteoporos Int. 2011 Dec;22(12):2963-72. doi: 10.1007/s00198-011-1533-1. Epub 2011 Feb 11. PMID 21311871
- [Result] Bessette L, Ste-Marie LG, Jean S, Davison KS, Beaulieu M, Baranci M, Bessant J, Brown JP. The care gap in diagnosis and treatment of women with a fragility fracture. Osteoporos Int. 2008 Jan;19(1):79-86. doi: 10.1007/s00198-007-0426-9. Epub 2007 Jul 20. PMID 17641811